CLINICAL TRIAL: NCT03930810
Title: NAtural Course and Prognosis of PFIC and Effect of Biliary Diversion (NAPPED Study), Meta-analysis of Individual Patient Data of PFIC Before and After Surgery (bile Diversion or Liver Transplantation)
Brief Title: NAtural Course and Prognosis of PFIC and Effect of Biliary Diversion
Acronym: NAPPED
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Henkjan J. Verkade, Principal Investigator, Professor of Pediatrics, University Medical Center Groningen
Other Study IDs: METc2017.106
Record Dates: First submitted 2019-04-19; First posted 2019-04-29 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Progressive Familial Intrahepatic Cholestasis
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FIC1 deficiency (PFIC1), BSEP deficiency (PFIC2), MDR3 deficiency (PFIC3) and other PFIC subtypes
  Interventions: Procedure: Surgical biliary diversion

INTERVENTIONS:
Procedure: Surgical biliary diversion — Surgical interruption of enterohepatic circulation

SUMMARY:
The natural course of PFIC syndromes and the effect of diversion techniques, have so far not been characterized in a rigorous manner within a larger population of patients. In fact, the clinical or biochemical parameters which most directly define and/or predict the success of reduced enterohepatic circulation (either by surgical diversion or medically) are still unclear.

The present project aims to:

1. Define the natural course of disease in patients with genetically defined FIC1 deficiency (PFIC1), BSEP deficiency (PFIC2), MDR3 deficiency (PFIC3) and other subtypes of the PFIC disease family (including e.g. Myo5B deficiency, TJP2 deficiency, a.o.), with respect to relevant biochemical and clinical parameters (and if available, histological). Included will be patients homozygous for a known, disease-causing mutation, patients compound homozygous for two disease-causing mutations or heterozygous for one disease-causing mutation in combination with the corresponding clinical phenotype .
2. Define the change in the natural course of disease in response to biliary diversion surgery and or liver transplantation, based on short- and long(er)-term changes in biochemical (if available, histological) and clinical parameters, including outcome measures. Follow up after transplantation will be limited, follow up after surgical biliary diversion will be as long as possible.
3. Assessment of biochemical variables as possible surrogate endpoints for clinical hard endpoints. If possible this allows for identification of low-risk to high-risk patients early during follow-up.
4. If patient numbers permit, to establish genotype-phenotype relationships for the most common genetic mutations causing the indicated diseases.

Based on this project it is anticipated that the investigators are able:

* to characterize the variation in natural course of disease (whether or not genotype dependent) to allow clinicians to rationally select a target population for assessing the effect of medical intervention, rather than surgical biliary diversion);
* to identify and qualify one or more biomarkers that independently predict either improved or poor clinical outcomes of surgical biliary diversion;
* to investigate if the identified biomarker(s) can be used as surrogate end point(s) for assessing and predicting outcomes with novel interventional strategies.

ELIGIBILITY:
Inclusion Criteria:

Clinical suspicion for FIC1-, BSEP- or MDR3-deficiency or of any other subtype of the PFIC family

Ages: 0 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The diagnosis of PFIC needs to be performed according to the international guidelines, based on (episodes with) the clinical symtpoms and identification of disease-causing mutations in the respective genes.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-01-26 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with liver transplantation | at 18 years of age, as well as >18 years of age (until 65 years of age)
  Underwent liver transplant
Number of participants that succumbed | at 18 years of age, as well as >18 years of age (until 65 years of age)
  Succumbed

SECONDARY OUTCOMES:
Number of participant undergoing a surgical biliary diversion | at 5, 10, 15 and 18 years of age, as well as >18 years of age (until 65 years of age)
  Underwent surgical biliary diversion

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Wessel DBE, Gonzales E, Hansen BE, Verkade HJ. Defining the natural history of rare genetic liver diseases: Lessons learned from the NAPPED initiative. Eur J Med Genet. 2021 Jul;64(7):104245. doi: 10.1016/j.ejmg.2021.104245. Epub 2021 May 13. PMID 33991701
- [Background] Felzen A, van Wessel DBE, Gonzales E, Thompson RJ, Jankowska I, Shneider BL, Sokal E, Grammatikopoulos T, Kadaristiana A, Jacquemin E, Spraul A, Lipinski P, Czubkowski P, Rock N, Shagrani M, Broering D, Nicastro E, Kelly D, Nebbia G, Arnell H, Fischler B, Hulscher JBF, Serranti D, Arikan C, Polat E, Debray D, Lacaille F, Goncalves C, Hierro L, Munoz Bartolo G, Mozer-Glassberg Y, Azaz A, Brecelj J, Dezsofi A, Calvo PL, Grabhorn E, Hartleif S, van der Woerd WJ, Kamath BM, Wang JS, Li L, Durmaz O, Kerkar N, Jorgensen MH, Fischer R, Jimenez-Rivera C, Alam S, Cananzi M, Laverdure N, Ferreira CT, Guerrero FO, Wang H, Sency V, Kim KM, Chen HL, de Carvalho E, Fabre A, Bernabeu JQ, Zellos A, Alonso EM, Sokol RJ, Suchy FJ, Loomes KM, McKiernan PJ, Rosenthal P, Turmelle Y, Horslen S, Schwarz K, Bezerra JA, Wang K, Hansen BE, Verkade HJ; NAtural course and Prognosis of PFIC and Effect of biliary Diversion (NAPPED) Consortium. Genotype-phenotype relationships of truncating mutations, p.E297G and p.D482G in bile salt export pump deficiency. JHEP Rep. 2022 Nov 16;5(2):100626. doi: 10.1016/j.jhepr.2022.100626. eCollection 2023 Feb. PMID 36687469
- [Background] Pawlikowska L, Strautnieks S, Jankowska I, Czubkowski P, Emerick K, Antoniou A, Wanty C, Fischler B, Jacquemin E, Wali S, Blanchard S, Nielsen IM, Bourke B, McQuaid S, Lacaille F, Byrne JA, van Eerde AM, Kolho KL, Klomp L, Houwen R, Bacchetti P, Lobritto S, Hupertz V, McClean P, Mieli-Vergani G, Shneider B, Nemeth A, Sokal E, Freimer NB, Knisely AS, Rosenthal P, Whitington PF, Pawlowska J, Thompson RJ, Bull LN. Differences in presentation and progression between severe FIC1 and BSEP deficiencies. J Hepatol. 2010 Jul;53(1):170-8. doi: 10.1016/j.jhep.2010.01.034. Epub 2010 Apr 13. PMID 20447715
- [Background] Strautnieks SS, Byrne JA, Pawlikowska L, Cebecauerova D, Rayner A, Dutton L, Meier Y, Antoniou A, Stieger B, Arnell H, Ozcay F, Al-Hussaini HF, Bassas AF, Verkade HJ, Fischler B, Nemeth A, Kotalova R, Shneider BL, Cielecka-Kuszyk J, McClean P, Whitington PF, Sokal E, Jirsa M, Wali SH, Jankowska I, Pawlowska J, Mieli-Vergani G, Knisely AS, Bull LN, Thompson RJ. Severe bile salt export pump deficiency: 82 different ABCB11 mutations in 109 families. Gastroenterology. 2008 Apr;134(4):1203-14. doi: 10.1053/j.gastro.2008.01.038. Epub 2008 Jan 18. PMID 18395098
- [Background] Bull LN, van Eijk MJ, Pawlikowska L, DeYoung JA, Juijn JA, Liao M, Klomp LW, Lomri N, Berger R, Scharschmidt BF, Knisely AS, Houwen RH, Freimer NB. A gene encoding a P-type ATPase mutated in two forms of hereditary cholestasis. Nat Genet. 1998 Mar;18(3):219-24. doi: 10.1038/ng0398-219. PMID 9500542
- [Background] Davit-Spraul A, Fabre M, Branchereau S, Baussan C, Gonzales E, Stieger B, Bernard O, Jacquemin E. ATP8B1 and ABCB11 analysis in 62 children with normal gamma-glutamyl transferase progressive familial intrahepatic cholestasis (PFIC): phenotypic differences between PFIC1 and PFIC2 and natural history. Hepatology. 2010 May;51(5):1645-55. doi: 10.1002/hep.23539. PMID 20232290
- [Background] Bull LN, Pawlikowska L, Strautnieks S, Jankowska I, Czubkowski P, Dodge JL, Emerick K, Wanty C, Wali S, Blanchard S, Lacaille F, Byrne JA, van Eerde AM, Kolho KL, Houwen R, Lobritto S, Hupertz V, McClean P, Mieli-Vergani G, Sokal E, Rosenthal P, Whitington PF, Pawlowska J, Thompson RJ. Outcomes of surgical management of familial intrahepatic cholestasis 1 and bile salt export protein deficiencies. Hepatol Commun. 2018 Mar 30;2(5):515-528. doi: 10.1002/hep4.1168. eCollection 2018 May. PMID 29761168
- [Background] Droge C, Bonus M, Baumann U, Klindt C, Lainka E, Kathemann S, Brinkert F, Grabhorn E, Pfister ED, Wenning D, Fichtner A, Gotthardt DN, Weiss KH, McKiernan P, Puri RD, Verma IC, Kluge S, Gohlke H, Schmitt L, Kubitz R, Haussinger D, Keitel V. Sequencing of FIC1, BSEP and MDR3 in a large cohort of patients with cholestasis revealed a high number of different genetic variants. J Hepatol. 2017 Dec;67(6):1253-1264. doi: 10.1016/j.jhep.2017.07.004. Epub 2017 Jul 19. PMID 28733223
- [Background] Wang KS, Tiao G, Bass LM, Hertel PM, Mogul D, Kerkar N, Clifton M, Azen C, Bull L, Rosenthal P, Stewart D, Superina R, Arnon R, Bozic M, Brandt ML, Dillon PA, Fecteau A, Iyer K, Kamath B, Karpen S, Karrer F, Loomes KM, Mack C, Mattei P, Miethke A, Soltys K, Turmelle YP, West K, Zagory J, Goodhue C, Shneider BL; Childhood Liver Disease Research Network (ChiLDReN). Analysis of surgical interruption of the enterohepatic circulation as a treatment for pediatric cholestasis. Hepatology. 2017 May;65(5):1645-1654. doi: 10.1002/hep.29019. Epub 2017 Mar 22. PMID 28027587
- [Background] van Wessel DBE, Thompson RJ, Gonzales E, Jankowska I, Sokal E, Grammatikopoulos T, Kadaristiana A, Jacquemin E, Spraul A, Lipinski P, Czubkowski P, Rock N, Shagrani M, Broering D, Algoufi T, Mazhar N, Nicastro E, Kelly DA, Nebbia G, Arnell H, Bjorn Fischler, Hulscher JBF, Serranti D, Arikan C, Polat E, Debray D, Lacaille F, Goncalves C, Hierro L, Munoz Bartolo G, Mozer-Glassberg Y, Azaz A, Brecelj J, Dezsofi A, Calvo PL, Grabhorn E, Sturm E, van der Woerd WJ, Kamath BM, Wang JS, Li L, Durmaz O, Onal Z, Bunt TMG, Hansen BE, Verkade HJ; NAtural course and Prognosis of PFIC and Effect of biliary Diversion (NAPPED) consortium. Genotype correlates with the natural history of severe bile salt export pump deficiency. J Hepatol. 2020 Jul;73(1):84-93. doi: 10.1016/j.jhep.2020.02.007. Epub 2020 Feb 20. PMID 32087350
- [Background] van Wessel DBE, Thompson RJ, Gonzales E, Jankowska I, Shneider BL, Sokal E, Grammatikopoulos T, Kadaristiana A, Jacquemin E, Spraul A, Lipinski P, Czubkowski P, Rock N, Shagrani M, Broering D, Algoufi T, Mazhar N, Nicastro E, Kelly D, Nebbia G, Arnell H, Fischler B, Hulscher JBF, Serranti D, Arikan C, Debray D, Lacaille F, Goncalves C, Hierro L, Munoz Bartolo G, Mozer-Glassberg Y, Azaz A, Brecelj J, Dezsofi A, Luigi Calvo P, Krebs-Schmitt D, Hartleif S, van der Woerd WL, Wang JS, Li LT, Durmaz O, Kerkar N, Horby Jorgensen M, Fischer R, Jimenez-Rivera C, Alam S, Cananzi M, Laverdure N, Targa Ferreira C, Ordonez F, Wang H, Sency V, Mo Kim K, Chen HL, Carvalho E, Fabre A, Quintero Bernabeu J, Alonso EM, Sokol RJ, Suchy FJ, Loomes KM, McKiernan PJ, Rosenthal P, Turmelle Y, Rao GS, Horslen S, Kamath BM, Rogalidou M, Karnsakul WW, Hansen B, Verkade HJ; Natural Course and Prognosis of PFIC and Effect of Biliary Diversion Consortium. Impact of Genotype, Serum Bile Acids, and Surgical Biliary Diversion on Native Liver Survival in FIC1 Deficiency. Hepatology. 2021 Aug;74(2):892-906. doi: 10.1002/hep.31787. Epub 2021 Jul 13. PMID 33666275